CLINICAL TRIAL: NCT01799694
Title: Phase II Clinical Trial to Study the Feasibility and Safety of the Expanded Autologous Stem Cells Use Derived From Adipose Tissue (e-ASC) for the Local Urinary Incontinence After a Radical Prostate Cancer Surgery
Brief Title: Stem Cells Treatment for the Local Urinary Incontinence After a Radical Prostate Cancer Surgery (HULPURO)
Acronym: FLPURO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLPURO-2009-01; 2009-016298-14 (EudraCT Number)
Record Dates: First submitted 2012-09-04; First posted 2013-02-27 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2012-09

CONDITIONS: Urinary Incontinence
Keywords: Urinary incontinence; Autologous expanded stem cells; Radical prostate cancer surgery
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Expanded Stem Cells (Experimental): Inject of Autologous Adipose-derived expanded stem cells
  Interventions: Drug: Inject of Autologous Adipose-derived stem cells

INTERVENTIONS:
Drug: Inject of Autologous Adipose-derived stem cells — Inject in muscle of autologous adipose derived stem cells
  Other Names: Autologuos eASC

SUMMARY:
The purpose of this study is to evaluate the feasibility and security of the autologous e-ASC for the urinary incontinence after a radical prostate cancer surgery

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Men over 18 years old. Good general state of health according to the findings of the clinical history and the physical examination
3. Prostate cancer diagnosed subjects via a biopsy and having had a radical surgery with a healing purpose in the previous 18 months
4. Having urinary incontinence after the surgery
5. Failure in any previous conservative treatment

Exclusion Criteria:

1. Having had an adjuvant treatment
2. Having a PSA ≥ 0,2 after surgery
3. Having any sign or symptom that suggest the investigator the non-healing of the adenocarcinoma
4. Active urine infection
5. Alcohol or other addictive substances abuse antecedents in the previous 6 months to the inclusion
6. Cardiopulmonary illness that, in the investigator opinion, could be unstable or could be serious enough to drop the patient from the study
7. Any kind of medical or psychiatric illness that, in the investigator opinion, could be a reason to exclude the patient from the study
8. Subjects with congenital or acquired immunodeficiencies, B and/or C Hepatitis, Tuberculose or Treponema diagnosed at the moment of inclusion
9. Anesthetic allergy
10. Major surgery or severe trauma in the previous 6 months
11. Administration of any drug under experimentation in the present or in the previous 3 months before recruitment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility and security of the autologous e-ASC for the urinary incontinence after a radical prostate cancer surgery | 16 weeks
  Possibility of inject ASc by cystoscope

SECONDARY OUTCOMES:
Quality of life assessment using the SF-12 Questionnaire | 1, 4, 16, 24 weeks
  SF-12 questionnaire
Adverse events | 1, 4, 16, 24 weeks
  Data collected

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Alonso Gregorio, MD, Principal Investigator — Cell Therapy laboratory and general Surgery Department, Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- [Background] Strasser H, Tiefenthaler M, Steinlechner M, Eder I, Bartsch G, Konwalinka G. Age dependent apoptosis and loss of rhabdosphincter cells. J Urol. 2000 Nov;164(5):1781-5. PMID 11025769
- [Background] Andriole GL, Grubb III LB, Buys SS et als. for the PLCO Project Team
- [Background] Schroder FH, Hugosson J, Roobol MJ, Tammela TL, Ciatto S, Nelen V, Kwiatkowski M, Lujan M, Lilja H, Zappa M, Denis LJ, Recker F, Berenguer A, Maattanen L, Bangma CH, Aus G, Villers A, Rebillard X, van der Kwast T, Blijenberg BG, Moss SM, de Koning HJ, Auvinen A; ERSPC Investigators. Screening and prostate-cancer mortality in a randomized European study. N Engl J Med. 2009 Mar 26;360(13):1320-8. doi: 10.1056/NEJMoa0810084. Epub 2009 Mar 18. PMID 19297566
- [Background] Mitterberger M, Pinggera GM, Marksteiner R, Margreiter E, Plattner R, Klima G, Strasser H. Functional and histological changes after myoblast injections in the porcine rhabdosphincter. Eur Urol. 2007 Dec;52(6):1736-43. doi: 10.1016/j.eururo.2007.05.007. Epub 2007 May 22. PMID 17532554
- [Background] Kwon D, Kim Y, Pruchnic R, Jankowski R, Usiene I, de Miguel F, Huard J, Chancellor MB. Periurethral cellular injection: comparison of muscle-derived progenitor cells and fibroblasts with regard to efficacy and tissue contractility in an animal model of stress urinary incontinence. Urology. 2006 Aug;68(2):449-54. doi: 10.1016/j.urology.2006.03.040. PMID 16904482
- [Background] Cannon TW, Lee JY, Somogyi G, Pruchnic R, Smith CP, Huard J, Chancellor MB. Improved sphincter contractility after allogenic muscle-derived progenitor cell injection into the denervated rat urethra. Urology. 2003 Nov;62(5):958-63. doi: 10.1016/s0090-4295(03)00679-4. PMID 14624934
- [Background] Praud C, Sebe P, Bierinx AS, Sebille A. Improvement of urethral sphincter deficiency in female rats following autologous skeletal muscle myoblasts grafting. Cell Transplant. 2007;16(7):741-9. doi: 10.3727/000000007783465118. PMID 18019363
- [Background] Becker C, Jakse G. Stem cells for regeneration of urological structures. Eur Urol. 2007 May;51(5):1217-28. doi: 10.1016/j.eururo.2007.01.029. Epub 2007 Jan 18. PMID 17254699
- [Background] Zuk PA, Zhu M, Mizuno H, Huang J, Futrell JW, Katz AJ, Benhaim P, Lorenz HP, Hedrick MH. Multilineage cells from human adipose tissue: implications for cell-based therapies. Tissue Eng. 2001 Apr;7(2):211-28. doi: 10.1089/107632701300062859. PMID 11304456
- [Background] Kajbafzadeh AM, Elmi A, Payabvash S, Salmasi AH, Saeedi P, Mohamadkhani A, Sadeghi Z, Nikfarjam L. Transurethral autologous myoblast injection for treatment of urinary incontinence in children with classic bladder exstrophy. J Urol. 2008 Sep;180(3):1098-105. doi: 10.1016/j.juro.2008.05.057. Epub 2008 Jul 18. PMID 18639289
- [Background] Carr LK, Steele D, Steele S, Wagner D, Pruchnic R, Jankowski R, Erickson J, Huard J, Chancellor MB. 1-year follow-up of autologous muscle-derived stem cell injection pilot study to treat stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Jun;19(6):881-3. doi: 10.1007/s00192-007-0553-z. PMID 18204978
- [Background] Mitterberger M, Marksteiner R, Margreiter E, Pinggera GM, Frauscher F, Ulmer H, Fussenegger M, Bartsch G, Strasser H. Myoblast and fibroblast therapy for post-prostatectomy urinary incontinence: 1-year followup of 63 patients. J Urol. 2008 Jan;179(1):226-31. doi: 10.1016/j.juro.2007.08.154. Epub 2007 Nov 14. PMID 18001790
- [Background] Mitterberger M, Pinggera GM, Marksteiner R, Margreiter E, Fussenegger M, Frauscher F, Ulmer H, Hering S, Bartsch G, Strasser H. Adult stem cell therapy of female stress urinary incontinence. Eur Urol. 2008 Jan;53(1):169-75. doi: 10.1016/j.eururo.2007.07.026. Epub 2007 Jul 23. PMID 17683852
- [Background] García Olmo D, García-Verdugo JM, Alemany J, Gonzalez M, Gutierrez-Fuentes JA. CELL THERAPHY . Ed. Mac Graw Hill. Madrid 2007
- [Background] Garcia-Olmo D, Garcia-Arranz M, Garcia LG, Cuellar ES, Blanco IF, Prianes LA, Montes JA, Pinto FL, Marcos DH, Garcia-Sancho L. Autologous stem cell transplantation for treatment of rectovaginal fistula in perianal Crohn's disease: a new cell-based therapy. Int J Colorectal Dis. 2003 Sep;18(5):451-4. doi: 10.1007/s00384-003-0490-3. Epub 2003 May 20. PMID 12756590
- [Background] Garcia-Olmo D, Herreros D, Pascual I, Pascual JA, Del-Valle E, Zorrilla J, De-La-Quintana P, Garcia-Arranz M, Pascual M. Expanded adipose-derived stem cells for the treatment of complex perianal fistula: a phase II clinical trial. Dis Colon Rectum. 2009 Jan;52(1):79-86. doi: 10.1007/DCR.0b013e3181973487. PMID 19273960